CLINICAL TRIAL: NCT05658263
Title: Bacterial Intestinal Gut Modification Around Cancer Surgery (BIG MACS) Diet
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SURG-2023-31051
Record Dates: First submitted 2022-10-11; First posted 2022-12-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Dysbiosis; Sarcopenia; Colon Cancer
MeSH Terms: conditions — Dysbiosis; Sarcopenia; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Diet (Active Comparator): Participants receiving only standard of care (SOC) nutrition advice, which is SOC Dietary Instructions, as provided by routine surgical consults and one protein shake per day for 4 weeks prior to surgery (SOC).
  Interventions: Dietary Supplement: Standard Diet
- BIG MACS Diet (Experimental): Participants will be instructed to consume the study diet, referred to as the 'BIG MACS Diet' and one protein shake per day for 4 weeks prior to surgery (SOC). Following surgery, participants will continue to follow the BIG MACS Diet for an additional four weeks, with solid food reintroduction after surgery as early as tolerated.
  Interventions: Dietary Supplement: BIG MACS Diet

INTERVENTIONS:
Dietary Supplement: Standard Diet — Participants receiving only standard of care (SOC) nutrition advice, which is SOC Dietary Instructions, as provided by routine surgical consults and one protein shake per day for 4 weeks prior to surgery (SOC).
  Arms: Standard Diet
Dietary Supplement: BIG MACS Diet — Participants will be instructed to consume the study diet, referred to as the 'BIG MACS Diet' and one protein shake per day for 4 weeks prior to surgery (SOC). Following surgery, participants will continue to follow the BIG MACS Diet for an additional four weeks, with solid food reintroduction after surgery as early as tolerated.
  Arms: BIG MACS Diet

SUMMARY:
The long-term study objective is to develop optimized nutritional therapies for surgery and test them in clinical practice. This pilot study will test a microbiome-optimization diet in colorectal cancer surgery patients. The study hypothesizes that the Bacterial Intestinal Gut Modification Around Cancer Surgery (BIG MACS) Diet will provide participants with increased microbiota accessible carbohydrates (MACs) to support the microbiome and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70 years
* Primary diagnosis of colon cancer, stages 1-3.
* Able and willing to provide informed consent.
* English-speaking.
* Willingness to return to the study site for specified study visits at D7 and D30.
* Able to comply with study measures.

Exclusion Criteria:

* Age ≤ 25 years or ≥70 years
* If surgery is being performed for any reason other than resection of colon cancer. Neoadjuvant therapy, or if surgery is not the initial approach for the patient's colon cancer treatment
* Significant anemia (hemoglobin 1.0 g/dL or more below normal range) or history of coagulopathy: any personal history of hereditary or acquired bleeding disorder, or thrombocytopenia with platelets under 100,000.
* Serum creatinine greater than 1.5 mg/dL.
* Serum total bilirubin greater than the upper limit of normal in the absence of Gilbert's syndrome or alkaline phosphatase or ALT or AST greater than 2.5 times the upper limit of normal. Elevated INR (1.5 or above).
* Alcohol intake more than one drink or greater than 20 grams per day for women or 30 grams per day for men.
* History of gastrointestinal surgery including stomach, small bowel or colon resection, pancreatic surgery, bile duct or gallbladder surgery, or splenectomy, or gastric bypass.
* History of intra-abdominal sepsis.
* Previous organ transplantation.
* Self-reported HIV-positive status, active tuberculosis, active malaria, chronic hepatitis B or C, cirrhosis, or inflammatory bowel disease.
* Currently pregnant or nursing.
* History of alcohol, drug, or opioid dependency (excluding nicotine) in the past five years.
* Active psychosocial or psychiatric problem that is likely to interfere with adherence to the protocol.
* Depression: A CES-D score more than 16 and a psychologist determining that the patient is not a good fit for surgery.
* Body mass index (BMI) <20 or > 40 kilograms per meter squared:

obesity is known to impact the microbiome and immune system and the occurrence of anastomotic leak, and extreme obesity may confound interpretation of these factors in association to leak. Inferences may be made by matching participants with less severe obesity (BMI <40).

* Presence of any type of non-MRI compatible implant, including cardiac pacemakers or defibrillators, neurostimulators, cochlear implants, or other metallic hardware
* Self-reported history of claustrophobia.
* Incarceration
* Inability to adhere to the study protocol, procedures, and diet
* Exclusions may also be made at the discretion of the attending physician.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | baseline and 4 weeks after surgery
  The change in muscle mass assessed by MRI-measured area and density of the psoas muscle at the level of the L3 vertebra with adjunct grip strength measurement.
Frequency of accidental gas leakage | 4 weeks after surgery
  this will be assessed in times per day or times per month
Frequency of accidental mucus leakage | 4 weeks after surgery
  this will be assessed in times per day or times per month
Frequency of accidental liquid stool leakage | 4 weeks after surgery
  this will be assessed in times per day or times per month
Frequency of bowel movements | 4 weeks after surgery
  this will be assessed in numbers per day or numbers per week
stool consistency | 4 weeks after surgery
  Bristol Stool Chart: Type 1 (hard lumps) through Type 7 (watery, no solid pieces, entirely liquid
Bowel emptying patterns | 4 weeks after surgery
  (includes constipation, diarrhea, urgency; range: always--> never)
Laxative/stool softener use | 4 weeks after surgery
  Yes/No
Laxative/stool softener use | 4 weeks after surgery
  times/day
Laxative/stool softener use | 4 weeks after surgery
  times/week
Laxative/stool softener use | 4 weeks after surgery
  times/month
Gastrointestinal comfort | 24 hours before surgery
  range: 0 (no problem) --> 4 (very strong discomfort)
Bowel emptying patterns | 24 hours before surgery
  includes constipation, diarrhea, urgency; range: 0 (never) --> 4 (always)
Laxative/stool softener use | 24 hours before surgery
  range; 0-4+ doses
Compliance with the dietary intervention or standard of care- Baseline veggie meter | baseline
  carotenoid score, triplicate measurement; range: 0 (lower estimated value)-800 (arbitrary units; higher estimated value correlates with greater carotenoid concentrations
Compliance with the dietary intervention or standard of care- Baseline veggie meter | postop day 7
  carotenoid score, triplicate measurement; range: 0 (lower estimated value)-800 (arbitrary units; higher estimated value correlates with greater carotenoid concentrations
Compliance with the dietary intervention or standard of care- Baseline veggie meter | postop day 30
  carotenoid score, triplicate measurement; range: 0 (lower estimated value)-800 (arbitrary units; higher estimated value correlates with greater carotenoid concentrations
Compliance with the dietary intervention or standard of care- survey | 4 weeks
  24-hour diet recall surveys conducted by Nutrition Coordinating Center at University of Minnesota

SECONDARY OUTCOMES:
Change in microbiome features- alpha diversity | Baseline, time of surgery, postop day 7 and 30
  Shannon, Simpson, and Chao1 indices
Change in microbiome features- beta diversity | Baseline, time of surgery, postop day 7 and 30
  compositionally corrected Aitchison's distances
Fecal metabolites | baseline and 4 weeks after surgery
  Targeted fecal and serum metabolomics will measure changes in short chain fatty acids (SCFAs) and bile acids.
Fecal inflammatory markers | Baseline and 4 weeks after surgery
  ELISA. Fecal calprotectin and IgA levels will be measured using ELISA as markers of intestinal inflammation.
Changes in body composition- abdominal muscle | Baseline, time of surgery, postop day 7 and 30
  total abdominal muscle area in cm squared. Absolute and relative change in total abdominal muscle area per patient over time (cm squared ), with the average change per patient group compared between study and control group
Changes in body composition- psoas muscle | Baseline, time of surgery, postop day 7 and 30
  total psoas muscle area in cm squared. Absolute and relative change in total psoas muscle area per patient over time (cm squared ), with the average change per patient group compared between study and control group
Changes in body composition- volume of fat | Baseline, time of surgery, postop day 7 and 30
  MRI-measured area (cm2) and volume (L) of subcutaneous and visceral adipose tissue
Changes in body composition- liver fat | Baseline, time of surgery, postop day 7 and 30
  MRI-measured liver fat content

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Jahansouz, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided